CLINICAL TRIAL: NCT02458755
Title: Intensive Statin Treatment in Acute Ischemic Stroke Patients With INtracranial Atherosclerosis - High-Resolution Magnetic Resonance Imaging Study (STAMINA-MRI Study)
Brief Title: Intensive Statin Treatment in Acute Ischemic Stroke Patients With INtracranial Atherosclerosis
Acronym: STAMINA-MRI
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Collaborators: Don-A Pharmaceutical, Seoul, South Korea (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SMC 2011-12-053
Record Dates: First submitted 2015-05-05; First posted 2015-06-01 (Estimated); Last update posted 2017-04-26 (Actual); Status verified 2016-10

CONDITIONS: Stroke; Intracranial Atherosclerosis
MeSH Terms: conditions — Stroke; Intracranial Arteriosclerosis | interventions — Rosuvastatin Calcium; Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- High-dose statin treatment (Experimental): Atorvastatin (40mg) or Rosuvastatin (20mg)
  Interventions: Drug: High-dose statin: Atorvastatin 40mg or Rosuvastatin 20mg

INTERVENTIONS:
Drug: High-dose statin: Atorvastatin 40mg or Rosuvastatin 20mg — Atorvastatin 40mg or Rosuvastatin 20mg
  Other Names: Atorvastatin 40mg or Rosuvastatin 20mg

SUMMARY:
Purpose: Intracranial atherosclerosis is a common condition in Korean population consisting over 25% of ischemic stroke etiology. American Stroke Association and Korean Stroke Society recommend antiplatelet and statin for the treatment of intracranial atherosclerosis. Besides lowering blood cholesterol levels statin also stabilize atherosclerotic plaque and eventually lower the risk of ischemic stroke. However, little evidence resides on the effect of statin treatment on intracranial atherosclerosis. Recent advance in high-tesla magnetic resonance imaging enables direct imaging of intracranial atherosclerotic plaque and further assessment of treatment efficacy of statin in stabilization of intracranial atherosclerotic plaque became possible.

ELIGIBILITY:
Inclusion Criteria:

* Acute ischemic stroke patients within 7 days of symptom onset
* Symptomatic intracranial artery stenosis (above 30%) at proximal portion of middle cerebral artery (MCA), basilar artery, or intracranial portion of intracranial artery (ICA).
* Not receiving statins (HMA-coA reductase)
* Willing and able to comply with scheduled visits, lifestyle guidelines, treatment plan, laboratory tests, and other study procedures.

Exclusion Criteria:

* Extracranial artery (carotid artery bifurcation, proximal vertebral artery) stenosis above 50%
* Stroke attributable to cardioembolic origin (atrial fibrillation, valvular heart disease, aortic arch atherosclerosis)
* Severe hepatic or renal dysfunction
* Pregnant females as determined by positive urine hCG test or lactating females
* Subjects considered unwilling or unable to comply with the imaging procedures and study visit schedule

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2012-02; Primary Completion 2018-06 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Changes in vascular remodeling before and after the statin treatment | During initial admission and 6 months from stroke onset
  Changes in vascular remodeling before and after the statin treatment: Difference of lumen area, vessel area, wall area, remodeling index, wall area index, plaque volume, plaque composition and enhancement pattern on high-resolution MRI

SECONDARY OUTCOMES:
Elevated liver function test or muscle enzyme levels | During initial admission, an expected average of 1 week, and 1 and 3 month after discharge
  Abnormal laboratory findings of elevated liver function test or muscle enzyme levels
Recurrent stroke/Transient ischemic attack | Admission to study completion date, an expected average of 1 year
All causes of death | Admission to study completion date, an expected average of 1 year
  All causes of death including vascular and non-vascular death
Exploration of biomarkers | During initial admission, an expected average of 1 week
  Lipid profile, lipoprotein(a), apoB/A1, extracellular vesicles, and genetic polymorphisms associated with statin response.

CONTACTS AND LOCATIONS:
Locations (1):
- Oh Young Bang, Seoul, South Korea

REFERENCES:
- [Derived] Sim JE, Song HN, Choi JU, Lee JE, Baek IY, Cho HH, Kim JH, Chung JW, Kim GM, Park HJ, Bang OY, Seo WK. The effect of intensive statin therapy in non-symptomatic intracranial arteries: The STAMINA-MRI sub-study. Front Neurol. 2023 Mar 28;14:1069502. doi: 10.3389/fneur.2023.1069502. eCollection 2023. PMID 37056360
- [Derived] Chung JW, Cha J, Lee MJ, Yu IW, Park MS, Seo WK, Kim ST, Bang OY. Intensive Statin Treatment in Acute Ischaemic Stroke Patients with Intracranial Atherosclerosis: a High-Resolution Magnetic Resonance Imaging study (STAMINA-MRI Study). J Neurol Neurosurg Psychiatry. 2020 Feb;91(2):204-211. doi: 10.1136/jnnp-2019-320893. Epub 2019 Aug 1. PMID 31371644